CLINICAL TRIAL: NCT04616157
Title: Internet-based Cognitive Behavioral Therapy for Adolescents With Sleep Problems- a Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Mats Lekander, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/2315-31/2
Record Dates: First submitted 2018-04-05; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Insomnia Disorder; Depressive Disorder; Anxiety Disorders; Pain, Chronic; Inflammation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder; Anxiety Disorders; Chronic Pain; Inflammation

STUDY DESIGN:
Intervention Model Description: All participants will receive treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICBT-I (Experimental): The ICBT-I treatment program is a web-based intervention consisting of six chapters/sessions that adolescents go through during six consecutive weeks.The program starts with psychoeducation regarding sleep disorders and the rationale for a cognitive behavioral intervention. The main focus for the treatment is behavioral interventions, mainly sleep restriction and stimulus control. The intervention also addresses problem solving, maintenance of treatment gains, relapse prevention and relaxation techniques. Caregivers will not actively participate in the treatment. During the treatment phase participants will be in contact with a therapist through standardized forms in the program.
  Interventions: Behavioral: ICBT-I

INTERVENTIONS:
Behavioral: ICBT-I — Cognitive-behavioral therapy for insomnia

SUMMARY:
The primary objective of this study is to test the feasibility and efficacy of Internet-delivered Cognitive Behavioral Therapy (CBT) for adolescents (13 - 17 years) with sleep problems (ICBT-I). All participants will receive ICBT-I for six weeks. The investigators will also evaluate the effect of the intervention on comorbid psychiatric symptoms and function.

DETAILED DESCRIPTION:
PARTICIPANT RECRUITMENT:

For recruitment, this pilot trial will be advertised at child and adolescent mental health services and primary care clinics, as well as through newspapers. The inclusion procedure will be carried out in two steps: 1) telephone interview and 2) face-to-face assessment.

Telephone interview: An initial telephone interview will be conducted with the adolescent/parent in order to broadly assess inclusion and exclusion criteria.

Face-to-face baseline diagnostic assessment: After the telephone screening, the adolescent along with his/her parents, are invited to a face-to-face assessment at the Child and Adolescent Mental Health clinic, including the diagnostic screening interview MINI-KID conducted with adolescents and parents jointly. Insomnia diagnoses will be established using DSM-IV criteria and levels of insomnia symptoms will be determined using ISI-a. If the ISI-a score is >10, the family will be invited to participate in the study, provided that the other inclusion criteria are fulfilled and no exclusion criteria prohibit participation. Following face-to-face assessment, participants will be provided with an information sheet and consent form.

DATA COLLECTION:

Baseline self-report measures: Participants included in the study after the face-to-face diagnostic assessment are asked to fill in self-report measures on the internet, provided via personal login and password. Participants will aslo be asked to fill in a sleep-wake diary and to wear an actigraph during seven consecutive days/nights.

Self-rating assessments during intervention: ISI-a is administered to adolescents every week during treatment.

Study participants are in regular contact (on a weekly basis) with experienced clinicians during the ICBT-I treatment. Clinicians that suspect any kind of adverse event during the assessment or treatment process will contact the parent via telephone as a first step of assessing the severity of the incident. Adverse events in this context are defined as an actual or potential situation that threatens the patient's well-being, e.g., suicide risk or an acute increase of symptoms. In the case of an adverse event, the clinician informs the study coordinator (LÅ) for a discussion of adequate action taking. If a continuation of the ICBT treatment is considered inappropriate with regard to the participants' best interest and well-being, the participant will be excluded from the study and parents/adolescents will be provided with proper referral information. Any adverse event will be reported in the planned publication of the pilot study.

Outcome measure reliability procedures: To ensure the reliability of the assessments conducted by study clinicians, all assessors will be trained by experienced instructors in the diagnostic screening instrument MINI-KID. All therapists that participate in the study will also be continuously trained in MINI-KID interviewing, assessment and diagnosing.

Post-treatment and follow-up measurement: Post-treatment measurement with actigraphy, sleep-wake diary and self-report measures will be conducted immediately after treatment (6 weeks after baseline). A follow-up measurement will be performed 6 months after treatment termination.

Referral of non-responders After the 6-month follow-up, all non-responders (defined as those participants who have not improved to a clinically meaningful degree according to ISI-a) will be referred to their local child-and adolescent psychiatric clinic for further treatment.

Statistical Analyses Outcomes will be described as significant changes in objective and subjective sleep and in clinician and self-rated measures of insomnia symptoms and comorbid symptoms, within-group effect sizes (Cohen's d), clinically significant improvement rates and remission rates. Analyses will involve t-tests as well as linear mixed-effects modeling. Randomness of missing data will be analyzed with logistic regression. Depending on the amount of missing data, multiple imputations will be employed to compensate for missing values.

ELIGIBILITY:
Inclusion Criteria:

* Clinical levels of insomnia symptoms, as determined by ISI-a >10.
* Age between 13 and 17 years
* Ability to read and write Swedish
* Daily access to the internet through a computer or similar device
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* Diagnosed with autism spectrum disorder, psychosis or bipolar disorder
* Present risk of suicide
* Ongoing substance dependence
* Completed CBT for sleep disorders within the last 6 months (defined as at least 5 sessions of CBT
* Ongoing use of central nervous system stimulant medication

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in insomnia symptom severity | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Insomnia Severity Index- adolescent version ISI is a seven-item measure that yields a quantitative index of sleep impairment and treatment outcome. Total scores range from 0 to 28, with higher scores indicating greater perceived insomnia severity. The instrument has been adapted to teenagers, ISI-a, and validated on Swedish teenagers.

SECONDARY OUTCOMES:
Change in subjective total sleep time | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Sleep Wake Diary (SWD). The SWD is a subjective measure of participants' sleeping and waking times, from which total sleep time expressed in minutes is derived.
Change in subjective sleep onset latency | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Sleep Wake Diary (SWD). The SWD is a subjective measure of participants' sleeping and waking times from which latency until falling asleep, expressed in minutes, is obtained.
Change in subjective wake after sleep onset | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Sleep Wake Diary (SWD). The SWD is a subjective measure of participants' sleeping and waking times in which time awake expressed in minutes after sleep onset is obtained.
Change in subjective sleep efficiency | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Sleep Wake Diary (SWD). The SWD is a subjective measure of participants' sleeping and waking times, from which sleep efficency is computed as the quota between time sleeping/time spent in bed, expressed in percentage. A higher percentage denotes longer time asleep.
Change in objective sleep total sleep time | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with wrist worn actigraph units. The actigraph unit will be worn during 7 consecutive days/nights at all three measurement occasion, from which total sleep time expressed in minutes is obtained.
Change in objective sleep onset latency | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with wrist worn actigraph units. The actigraph unit will be worn during 7 consecutive days/nights at all three measurement occasions, from which time in minutes before falling asleep is obtained.
Change in objective wake after sleep onset | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with wrist worn actigraph units. The actigraph unit will be worn during 7 consecutive days/nights at all three measurement occasions from which time being awake after sleep onset is obtained.
Change in objective sleep efficiency | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with wrist worn actigraph units. The actigraph unit will be worn during 7 consecutive days/nights at all three measurement occasions, from which sleep efficency is computed as the quota between time sleeping/time spent in bed, expressed in percentage. A higher percentage denotes longer time asleep.
Change in symptoms of insomnia | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Athens Insomnia Scale (AIS), a self-administered questionnaire consisting of eight items to measure symptoms of insomnia. Total scores range from 0 to 24. Higher scores indicate that responders more severe insomnia symptoms.
Change in symptoms of depression | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Center for Epidemiological Studies Depression Scale for Children (CES-DC). CES-DS is a 20-item self-report depression inventory that is widely used in research and has been validated on children and adolescents. Scores range from 0 to 60, in which higher scores suggest a greater presence of depressive symptoms.
Change in symptoms of depression 2 | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Revised Children's Anxiety and Depression Scale Child and Parent version (RCADS-C/P). RCADS-C/P is a child and parent self-report measure of anxiety and depression related psychopathology. The 48 items of the RCADS measures five domains of anxiety: generalized anxiety, panic anxiety, separation anxiety, social anxiety and obsessive-compulsive anxiety, as well as symptoms of depression. For depression, values range from 0 to 30, with higher values denoting more depressive symptoms.
Change in symptoms of generalized anxiety | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with RCADS-C/P (see above). RCADS-C/P is a child and parent self-report measure of anxiety and depression related psychopathology. The 48 items of the RCADS measures five domains of anxiety: generalized anxiety, panic anxiety, separation anxiety, social anxiety and obsessive-compulsive anxiety, as well as symptoms of depression. For generalized anxiety, scores range from 0 to 18, with higher values denoting more severe symptoms of anxiety.
Change in difficulties in emotion regulation | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Difficulties in Emotion Regulation Scale, short version (DERS-16), a self-rated questionnaire assessing difficulties to regulate emotion. DERS-16 can range from 16 to 80, with Higher scores reflect greater impairment.
Change in intensity of pain | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  A Visual Analogue Scale (VAS) will be used to measure intensity of participants' current and past pain.
  The scale consists of a line where the ends are defined as extreme limits (0 = no pain; 10 = worst possible pain) of pain experience
Change in daytime functioning | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Functional Disability Inventory (FDI), a 15-item self-rated questionnaire to measure level of day-time functioning. Scores range from 0 (no disability) to 60 (severe disability).
Change in daytime sleepiness 1 | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with Pediatric Daytime Sleepiness Scale (PDSS), a self-report scale consisting of 8 items. Scores range from 0-32, with higher scores indicating more daytime sleepiness.
Change in daytime sleepiness 2 | Change from before treatment to after (+6 weeks) and to 6 month after treatment
  Measured with the Karolinska Sleepiness Scale (KSS), a 9-point Likert scale, ranging from 1 to 9, with higher numbers denoting more sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Lekander, PhD, Study Chair — Karolinska Institutet
Locations (1):
- BUP KFE, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided